CLINICAL TRIAL: NCT00544986
Title: A Prospective,Open-label Study of Anastrozole in Post-menopausal Women With Hormone Sensitive Advanced Breast Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5391L00001
Record Dates: First submitted 2007-10-08; First posted 2007-10-16 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; post menopausal women; Post menopausal women with hormone sensitive advanced breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Anastrozole

SUMMARY:
The overall objective of the clinical study is to assess the tolerability and clinical efficacy of anastrozole in post-menopausal women with hormone sensitive advanced breast cancer in India.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be adult (age ≥ 18 years age) post-menopausal* women
2. Patients must be diagnosed with advanced breast cancer (histologically or cytological confirmation required) i.e. TNM stage III or IV disease (locally advanced or metastatic breast cancer) or locoregional recurrent disease, not suitable for treatment by local surgery or radiation therapy
3. Measurable or evaluable disease
4. Patients with ER/PR positive tumour or ER/PR unknown status
5. Patients must be suitable for endocrine treatment with anastrozole
6. Prior adjuvant chemotherapy or endocrine therapy for early breast cancer is allowed, provided such treatment was completed at least twelve months prior to study enrollment
7. Performance status 0-2 (As per WHO Classification)
8. Concurrent use of bisphosphonates is permitted.
9. Patients must give their written informed consent for participation in the study

Exclusion Criteria:

1. Patients with tumors known to be estrogen and progesterone receptor-negative.
2. Estrogen hormone replacement therapy, concurrently or within 6 weeks before randomization
3. Extensive visceral involvement (significant hepatic involvement, brain metastasis or pulmonary involvement > 50% of the lungs); serum liver enzymes SGOT and SGPT should be no greater than five times the upper limit of the reference range
4. Patients received bone marrow transplantation before randomization
5. Any concurrent medical illness (uncontrolled cardiac disease or diabetes mellitus) or laboratory abnormalities that would compromise safety or prevent interpretation of results
6. An estimated survival of less than 3 months from the start of Study drug treatment based on clinical judgment.
7. Any systemic investigational drug within the thirty days of enrollment into study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2005-06; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
1. Tolerability(safety) 2.Efficacy (a) Time to tumor progression TTP (b) Objective Response (OR) Rate (c) Symptom Evaluation

SECONDARY OUTCOMES:
Efficacy (a) Time to treatment failure TTF (b)Duration of Response DOR (c) Duration of Clinical Benefit

CONTACTS AND LOCATIONS:
Overall Officials: Poonamalle P Bapsy, MD, Principal Investigator — Kidwai Memorial Institute of Oncology, Bangalore, INDIA